CLINICAL TRIAL: NCT03667599
Title: A Randomized Phase 2 Study of Home Care Following Autologous Hematopoietic Stem Cell Transplantation
Brief Title: A Phase 2 Study of Home Care Following Autologous Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00089697
Record Dates: First submitted 2018-07-03; First posted 2018-09-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Well-being of Caregivers (Caregiver Strain Index)
MeSH Terms: interventions — Home Care Services

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home care (Experimental): This is the arm for patients who receive their transplant care in their homes.
  Interventions: Other: home care
- Hospital Care (No Intervention): Standard of care for stem cell transplant recipients where the aftercare is done in hospital.
- Clinic Care (No Intervention): Standard of care for stem cell transplant recipients who live at home but receive aftercare in the daily outpatient clinic.

INTERVENTIONS:
Other: home care — This is the interventional arm where patients receive the transplant care in their homes.
  Arms: Home care

SUMMARY:
This is a research study to compare the well-being (caregiver strain index) of caregivers of patients receiving home vs standard care after autologous hematopoietic stem cell transplant.

ELIGIBILITY:
Patient Inclusion Criteria:

* Scheduled to undergo an autologous hematopoietic stem cell transplant for any cancer or non-cancer illness
* Age 18-80 years
* Karnofsky Performance Scale KPS> 80
* Able to read/write English
* A home that is deemed, upon inspection, in suitable condition to serve as a medical home, within a 90-minute driving distance of Duke

Patient Exclusion Criteria:

* Lack of a caregiver
* Pregnant women
* Patients with a documented active infection prior to starting their preparative regimen. This includes grade 3 or higher viral, bacterial, or fungal infection.
* Use of homeopathic medications, prebiotics, or probiotics that may impact gut microbiota

Caregiver Inclusion Criteria:

* Identified by patient as their primary caregiver
* Meet standard clinical criteria for being a caregiver (able to drive and take care of patient)
* Age 18-80 years

Caregiver Exclusion Criteria:

None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-09-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Caregivers (Caregiver Strain Index) | 14 days
  To compare the quality of life (Caregiver Strain Index) in caregivers of patients receiving home vs standard care after autologous hematopoietic stem cell transplant.

SECONDARY OUTCOMES:
Measuring Caregiver Burden as recorded in a Time Diary | 1 year
Measuring Caregiver Self-Efficacy assessed by the Modified Lorig | 1 year
Measuring Caregiver Satisfaction assessed by Caregiver Satisfaction | 1 year
Measuring Caregiver Quality of Life as assessed by the FACT-GP | 1 year
Measuring Caregiver Quality of Life as assessed by the PROMIS-Global Health | 1 year
Measuring Caregiver Fatigue as assessed by the PROMIS-Fatigue | 1 year
Measuring Caregiver Fatigue as assessed by the PROMIS-Sleep | 1 year
Measuring Caregiver Mental Health as assessed by the PROMIS-Depression | 1 year
Measuring Caregiver Mental Health as assessed by the PROMIS-Anxiety | 1 year
Measuring Return to Work in Caregivers (Work Assessment) | 1 year
Overall Survival | 1 year
Disease Free Survival | 1 year
Rates of Overall Infections | 1 year
Rates of Bacterial Infections | 1 year
Rates of Viral Infections | 1 year
Rates of Fungal Infections | 1 year
Rates of Hospital Admission | 1 year
Transplant Length of Stay | 1 year
Measuring Quality of Life as assessed by the EQ-5D-5L | 1 year
Measuring Symptoms as assessed by MDASI scale | 1 year
Measuring Self-Efficacy as assessed by the Lorig | 1 year
Measuring Fatigue as assessed by the PROMIS-Fatigue | 1 year
Measuring Fatigue as assessed by the PROMIS-Sleep | 1 year
Measuring Mental Health as assessed by the PROMIS-Anxiety | 1 year
Measuring Mental Health as assessed by the PROMIS-Depression | 1 year
Measuring Out-of-Pocket Costs as recorded in a Cost Diary | 1 year
Measuring Return to Work as assessed by the Work Assessment | 1 year
Measuring Social Support as assessed by the PROMIS-Social Isolation | 1 year
Measuring Nutrition as assessed by the PG-SGA | 30 days
Measuring Hand Grip Strength | 1 year
Measuring Exercise as assessed by 6 minute walk test | 1 year
Measuring Changes in fecal samples as measured by 16s rRNA sequencing | 1 year
Measuring Changes in the skin flora (microbiome) | 1 year
Measuring treatment related mortality (TRM) | 1 year
Measuring adverse events as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | 1 year
Measuring Direct Medical Costs | 6 months
Measuring Health Resource Utilization using Duke University Health System (DUHS) records | 1 year
Measuring Indirect Costs (Patient's and Caregivers' Time) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Sung, MD, Principal Investigator — Duke Health; Nelson Chao, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States